CLINICAL TRIAL: NCT03816605
Title: Effects of Fibroblast Growth Factors 19 on the Expression of Insulin Receptor Substrate-1/Glucose Transporter-1 in Trophoblast Cells Cultured in High Glucose
Brief Title: FGF19 and the Expression of IRS-1 and GLUT-1 in Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Dongyu Wang, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: FGF19
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Gestational Diabetes Mellitus
Keywords: GDM; IRS-1; GLUT-1
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- control: Cells were cultured in the basic medium containing 2× penicillin and streptomycin antibody.
- Recombinant FGF19: Cells were cultured in the basic medium with recombinant FGF19 at concentration of 100ng/ml.
- High-glucose: Cells were cultured in the high-glucose medium at concentration of 25mM.
- FGF19 and HG: Cells were cultured in the medium with both recombinant FGF19 and high-glucose.

SUMMARY:
Insulin resistance plays a key role in the development of gestational diabetes mellitus(GDM). As the largest endocrine organ and the transport intermediary of maternal-fetal nutrient and a large of hormone and enzymes, placenta not only plays an important role in insulin resistance, but also have a profound effect on fetal growth and development.

Insulin receptor substrate(IRS)-1, as a key signaling protein, plays vital role in the downstream of insulin receptor signaling pathway. Many studies have suggested that the central part of insulin resistance may be the insulin receptor substrate defect and the abnormal expression of the gene or protein of IRS-1 is one of the molecular mechanisms of the dysfunction of the insulin signaling pathway. The expression of IRS-1 and its tyrosine phosphorylated protein decreased abnormally in placenta, skeletal muscle and adipose tissue of GDM patients, which might be a significant cause to insulin resistance in GDM.

Besides, glucose transporter-1(GLUT-1), which may play a major role in the glucose transporter in the placenta. The increase of blood glucose in patients with GDM has apparent up-regulating effect on the expression of GLUT-1 in the placenta, which is associated the development of offspring.

The investigators' previous study showed that FGF19 in serum, placenta and musculus rectus abdominis was significantly decreased in patients with GDM, and was related to insulin resistance. Thus, the investigators speculate that the abnormal expression of FGF19 may be involved in the development of insulin resistance in GDM patients and disorder of carbohydrate and lipid metabolism.

In the present study, the investigators will further investigate the effect of FGF19 on the expression of IRS-1/GLUT-1 in cultured trophoblast cells of high glucose, and probe into the effect of FGF19 on the insulin resistance and glucose transport.

DETAILED DESCRIPTION:
Women who choose to terminate pregnancy because of maternal factors at the first and second trimester, or delivered at term in the First Affiliated Hospital of Sun Yat-sen University were enrolled in the study.

Samples for measurement were obtained from women undergoing induced abortion or caesarean section. The villous trophoblast extracted from the placental villus were treated with recombinant FGF19, high glucose medium or both recombinant FGF19 and high glucose medium or neither. By the end of culture, mRNA and protein expression levels of IRS-1/GLUT-1 were investigated with real-time quantitative polymerase chain reaction (qRT-PCR) and western-blot, respectively. Clinical data were collected and analyzed.

Data were analyzed by SPSS20.0 database. The results were expressed as mean ± standard deviations, median or rate. Differences between groups were assessed by Student's unpaired t test, Mann-Whitney U test, or Chi-square test as appropriate. P values of <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Women who choose to terminate pregnancy because of maternal factors in the First Affiliated Hospital of Sun Yat-sen University at the 6-10 weeks of gestation.

Exclusion Criteria:

* Younger than 18 years old;
* Older than 40 years old;
* Diagnosed DM before pregnancy;
* Complicated with other diseases such as GDM, insulin resistance, obesity and related endocrine diseases, etc.;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University hospital
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Expression of IRS-1 and GLUT-1 in different group | six months
  concentration of IRS-1 and GLUT-1 in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Zilian Wang, M.D.,PhD, Study Director — O&G Department of the 1st affiliated hospital of Sun Yat-sen University
Locations (1):
- Obstetrics and Gynechology Department of the 1st affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China